CLINICAL TRIAL: NCT01013844
Title: Partner Assistance in Learning and Performing Skin Self-Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Loyola University (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003-01
Record Dates: First submitted 2009-11-11; First posted 2009-11-16 (Estimated); Results first posted 2011-03-10 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Melanoma
Keywords: skin self-examination; SSE; melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solo Learning (Active Comparator): Participant learning alone (without partner).
  Interventions: Behavioral: Skin Self Examination Information and ABCDE Rule
- Dyadic Learning (Active Comparator): Participant and partner learning together.
  Interventions: Behavioral: Skin Self Examination Information and ABCDE Rule

INTERVENTIONS:
Behavioral: Skin Self Examination Information and ABCDE Rule — Card with condensed information about skin self examination (SSE) and color illustrations of the ABCDE (asymmetry of shape, border irregularity, color variation, diameter > or equal to 6 mm, and evolution of the lesion) rule. A research assistant gave a skill demonstration using a magnifying lens.

SUMMARY:
This study is a behavioral science study designed to identify aspects of the dyadic relationship that promote Skin Self-Examination (SSE) in patients at high risk of developing melanoma. The patient is randomized to receive the educational intervention either as a solo learner or with the partner.

ELIGIBILITY:
Inclusion Criteria:

* Personal or family history of melanoma. If a personal history of melanoma, the patient was treated at least 1 month ago
* Evidence of dysplastic nevus syndrome or a large number of moles (Greater than 50)
* Able to see to read a newspaper, can read at an eighth grade level
* Speaks English
* 18 to 70 years old with a spouse or cohabitating partner

Exclusion Criteria:

* Under 18 years of age
* Patient overburden by other co-morbid diseases such as chronic immunosuppression from organ transplantation
* Have insufficient vision to to read a newspaper
* Unable to read English
* Have insufficient cognitive skills to follow instructions provided at an eighth grade language level

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P West, PhD, Study Director — Northwestern University; June K Robinson, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Background] Robinson JK, Stapleton J, Turrisi R. Relationship and partner moderator variables increase self-efficacy of performing skin self-examination. J Am Acad Dermatol. 2008 May;58(5):755-62. doi: 10.1016/j.jaad.2007.12.027. Epub 2008 Feb 6. PMID 18258332
- [Result] Robinson JK, Turrisi R. Skills training to learn discrimination of ABCDE criteria by those at risk of developing melanoma. Arch Dermatol. 2006 Apr;142(4):447-52. doi: 10.1001/archderm.142.4.447. PMID 16618863
- [Result] Robinson JK, Turrisi R, Stapleton J. Efficacy of a partner assistance intervention designed to increase skin self-examination performance. Arch Dermatol. 2007 Jan;143(1):37-41. doi: 10.1001/archderm.143.1.37. PMID 17224540
- [Result] Robinson JK, Turrisi R, Stapleton J. Examination of mediating variables in a partner assistance intervention designed to increase performance of skin self-examination. J Am Acad Dermatol. 2007 Mar;56(3):391-7. doi: 10.1016/j.jaad.2006.10.028. Epub 2006 Dec 4. PMID 17147966
- [Result] Glanz K, Yaroch AL, Dancel M, Saraiya M, Crane LA, Buller DB, Manne S, O'Riordan DL, Heckman CJ, Hay J, Robinson JK. Measures of sun exposure and sun protection practices for behavioral and epidemiologic research. Arch Dermatol. 2008 Feb;144(2):217-22. doi: 10.1001/archdermatol.2007.46. PMID 18283179
- [Result] Robinson JK, Ortiz S. Use of photographs illustrating ABCDE criteria in skin self-examination. Arch Dermatol. 2009 Mar;145(3):332-3. doi: 10.1001/archdermatol.2008.604. No abstract available. PMID 19289774
- [Result] Boone SL, Stapleton J, Turrisi R, Ortiz S, Robinson JK, Mallett KA. Thoroughness of skin examination by melanoma patients: influence of age, sex and partner. Australas J Dermatol. 2009 Aug;50(3):176-80. doi: 10.1111/j.1440-0960.2009.00533.x. PMID 19659978
- [Result] Robinson JK, Mallett KA, Turrisi R, Stapleton J. Engaging patients and their partners in preventive health behaviors: the physician factor. Arch Dermatol. 2009 Apr;145(4):469-73. doi: 10.1001/archdermatol.2009.2. No abstract available. PMID 19380671
- [Result] Robinson JK, Mallett KA. The duty to inspect the skin and counsel those at risk to develop melanoma. JAMA. 2009 Apr 22;301(16):1702-4. doi: 10.1001/jama.2009.542. No abstract available. PMID 19388140
- [Result] Robinson JK, Turrisi R, Mallett K, Stapleton J, Pion M. Comparing the efficacy of an in-person intervention with a skin self-examination workbook. Arch Dermatol. 2010 Jan;146(1):91-4. doi: 10.1001/archdermatol.2009.350. No abstract available. PMID 20083705
- [Derived] Robinson JK, Gaber R, Hultgren B, Eilers S, Blatt H, Stapleton J, Mallett K, Turrisi R, Duffecy J, Begale M, Martini M, Bilimoria K, Wayne J. Skin self-examination education for early detection of melanoma: a randomized controlled trial of Internet, workbook, and in-person interventions. J Med Internet Res. 2014 Jan 13;16(1):e7. doi: 10.2196/jmir.2883. PMID 24418949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from hospital registries of patients who were diagnosed as having cutaneous melanoma (CM) and were being seen at least annually by physicians for their skin conditions.
Period: Overall Study
Arm/Group | Solo Learning | Dyadic Learning
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solo Learning | Dyadic Learning | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 69 years | 54 | 61 | 115
  >=70 years | 11 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 33 | 32 | 65
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Skin Examinations Without Partner Over 4 Months
Description: Behavioral outcome was measured by assessing the number of times that participants examined their skin in the last 4 months.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Times examined skin by self
Groups:
- Solo Learning Baseline; Solo Learning Immediate Follow-up; Solo Learning 4-Month Follow-up: Participant learning alone (without partner).
- Dyadic Learning Baseline; Dyadic Learning Immediate Follow-up; Dyadic Learning 4-Month Follow-up: Participant and partner learning together.
Arm/Group | Solo Learning Baseline | Dyadic Learning Baseline | Solo Learning Immediate Follow-up | Dyadic Learning Immediate Follow-up | Solo Learning 4-Month Follow-up | Dyadic Learning 4-Month Follow-up
Number analyzed (Participants) | 65 | 65 | 65 | 65 | 65 | 65
Times examined skin by self | 0.02 (0.12) | 0.00 (0.00) | 0.02 (0.12) | 0.00 (0.00) | 0.23 (0.42) | 0.80 (0.74)

2. Primary Outcome: Mean Number of Skin Examinations With Partner Over 4 Months
Description: Behavioral outcome was measured by assessing the number of times that participants examined their skin with a partner in the last 4 months.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Times examined skin with a partner
Arm/Group | Solo Learning Baseline | Dyadic Learning Baseline | Solo Learning Immediate Follow-up | Dyadic Learning Immediate Follow-up | Solo Learning 4-Month Follow-up | Dyadic Learning 4-Month Follow-up
Number analyzed (Participants) | 65 | 65 | 65 | 65 | 65 | 65
Times examined skin with a partner | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.23 (0.42) | 0.81 (0.72)

3. Primary Outcome: Mean Number of Times Reviewed Skin Self Examination Guidelines Over 4 Months
Description: Behavioral outcome was measured by assessing the number of times that participants reviewed skin self examination guidelines in the last 4 months.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Number of times reviewed SSE guidelines
Arm/Group | Solo Learning Baseline | Dyadic Learning Baseline | Solo Learning Immediate Follow-up | Dyadic Learning Immediate Follow-up | Solo Learning 4-Month Follow-up | Dyadic Learning 4-Month Follow-up
Number analyzed (Participants) | 65 | 65 | 65 | 65 | 65 | 65
Number of times reviewed SSE guidelines | .03 (0.17) | 0.0 (0.0) | 0.08 (0.27) | 0.0 (0.0) | 0.55 (0.53) | 0.91 (0.68)

ADVERSE EVENTS:
Time Frame: 4 months
Description: 130 subjects were enrolled in the study and 130 subjects were at risk.
Arm/Group | Solo Learning | Dyadic Learning
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No